CLINICAL TRIAL: NCT04309968
Title: A Phase I Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Anti-tumor Activity of SYHA1801 Capsules in Patients With Advanced Solid Tumors.
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK) and Anti-tumor Activity of SYHA1801 Monotherapy in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYHA1801201901/PRO
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- solid tumors (Experimental): Experimental: Solid tumors Part 1 - Dose-escalation of SYHA1801 in patients with advanced solid tumors.Daily dosing of SYHA1801 on Days 1 and 4-31 of 28-day cycle. Escalating dose cohorts.
  Interventions: Drug: Drug: SYHA1801
- advanced cancers (Experimental): Part 2 - Dose-expansion of SYHA1801 in patients with advanced cancers potentially sensitive to BRD4 inhibitor.The dose level and schedule of SYHA1801 of 28-day cycle at the MTD determined in Part 1.
  Interventions: Drug: Drug: SYHA1801

INTERVENTIONS:
Drug: Drug: SYHA1801 — Drug: SYHA1801 administered orally

SUMMARY:
This is a safety, pharmacokinetic and pharmacodynamic study designed to estimate the maximum tolerated dose (MTD), and determine the Recommended Phase 2 Dose (RP2D) of SYHA1801, a BRD4 inhibitor in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study will be performed in two parts. Part 1 will enroll patients with advanced solid tumors. Patients will receive SYHA1801 orally on Days 1 and 4-31 in the first cycle. Enrollment will follow a dose-escalation schedule until grade 3 drug-related adverse events are observed, at this point the i3+3 enrollment design will be used. Dose increments will be guided by data generated from previous levels. The dose and possibly the schedule will be adjusted to determine the Maximum Tolerated Dose (MTD). If a patient wishes to continuously receive study treatment on completion of Cycle 1, the patient can continue study treatment in 28-day Cycle 2 and subsequent cycles.

Part 2 will enroll patients with specific solid tumor which might potentially respond to BRD4 inhibitor. Patients will receive SYHA1801 at a dose and schedule established in Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, ≤75 years, no gender limitation.
2. Histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumors, for which standard therapy either does not exist or has proven ineffective, intolerable or inacceptable for the patient.
3. At least one measurable lesion as per RECIST version 1.1.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤1.
5. Life expectancy ≥3 months.
6. Adequate bone marrow reserve, renal and liver function.
7. Women of childbearing potential should agree to use contraceptive measures (such as IUD, contraceptive or condom) during the study and within 6 months after the end of the study; the serum pregnancy test should be negative within 7 days before enrollment, and must be non-lactating subjects; men should agree to use contraceptive measures during the study and within 6 months after the end of the study.
8. Signed informed consent form.

Exclusion Criteria:

1. Administration of chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy and other anti-tumor treatment within 4 weeks before the first dose of the study drug, except the following: using nitrosourea and mitomycin C within 6 weeks, using fluorouracil and small molecule targeted drugs within 2 weeks (or within 5 half time period), using traditional Chinese medicine with anti-tumor indications within 2 weeks.
2. Administration of other unlisted clinical research drugs within 4 weeks before the first dose of SYHA1801.
3. Major organ surgery (excluding biopsy) or significant trauma within 4 weeks before the first dose of SYHA1801.
4. Administration of glucocorticoids or other immunosuppressants within 14 days prior to the first dose of SYHA1801, except the following: local, ocular, intraarticular, intranasal and inhaled glucocorticoids; short-term use of glucocorticoids for preventive treatment.
5. Concomitant therapy with strong CYP3A4 inhibitors or inducers within 14 days.
6. Prior treatment with BET inhibitors.
7. Persistent grade >1 clinically significant toxicity related to prior antineoplastic therapies (except alopecia).
8. Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence that the patient's central nervous system metastasis or meningeal metastasis has not been controlled, that is not suitable for the group according to the judgment of the investigator.
9. Uncontrollable active infection.
10. History of autoimmune diseases, immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency, or organ transplant history.
11. Active hepatitis B; positive for hepatitis C antibody.
12. History of serious cardiovascular disease.
13. Inability to swallow oral medications or presence of a gastrointestinal disorder deemed to jeopardize intestinal absorption of SYHA1801.
14. Other serious illness or medical conditions.
15. Alcohol or drug dependence.
16. A clear history of neurological or psychiatric disorders.
17. Pregnant or breast-feeding female.
18. In the opinion of the investigator, not suitable for enrollment due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate AE,SAE and DLT of SYHA1801. | 28 days
  The occurrence and frequency of AE, SAE and DLT. To evaluate the safety and tolerability of SYHA1801.
To evaluate the MTD of SYHA1801 | through study completion, an average of 1 year
  The maximum tolerable dose (MTD) (if it has), recommended phase II dose (RP2D) and dosage regimen of SYHA1801.

SECONDARY OUTCOMES:
AUC0-last of SYHA1801. | 31 days
  To evaluate AUC0-last of SYHA1801.
AUC0-∞ of SYHA1801. | 31 days
  To evaluate AUC0-∞ of SYHA1801.
Cmax of SYHA1801. | 31 days
  To evaluate Cmax of SYHA1801.
Tmax of SYHA1801. | 31 days
  To evaluate Tmax of SYHA1801.
t½ of SYHA1801. | 31 days
  To evaluate t½ of SYHA1801.
CL/F of SYHA1801. | 31 days
  To evaluate CL/F of SYHA1801.
ORR of SYHA1801 | 2 months
  To evaluate ORR of SYHA1801
PFS of SYHA1801 | 2 months
  To evaluate PFS of SYHA1801
DCR of SYHA1801 | 2 months
  To evaluate DCR of SYHA1801
DOR of SYHA1801 | 2 months
  To evaluate DOR of SYHA1801

OTHER OUTCOMES:
Biomarkers and Beneficiaries | 2 months
  To evaluate potential pharmacodynamic biomarkers（C-MYC、MYCN、BCL-2、HEXIM1、CCR2、CD180、VEGFA） and to assess potential beneficiaries（such as hematoma tumors and myelofibrosis）

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China